CLINICAL TRIAL: NCT00690508
Title: Validation of Supra-Sternal Tube-Tip Palpation (SSTTP): A Method to Identify Correct Depth of Intubation in Infants and Children
Brief Title: Validation of Supra-Sternal Tube-Tip Palpation
Acronym: SSTTP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ottawa (Other)
Responsible Party: Uwe Schwarz, M.D., Dr. med, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 07/35X
Record Dates: First submitted 2008-04-07; First posted 2008-06-04 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Tracheal Intubation
Keywords: Intubation, Trachea, Sternum,; Tube tip, Tube placement, Tube tip palpation,; Validate; use; SSTTP; corrrect; placement
MeSH Terms: conditions — Tracheal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Supra-Sternal Tube-Tip Palpation (SSTTP) — The supra-sternal palpation of the tube after tracheal intubation.

SUMMARY:
Background:

The intra-tracheal intubation of a patient is a most delicate medical procedure performed under often life-threatening conditions in in- and out-of-hospital acute care medicine. Correct placement of the tube after intra-tracheal intubation is thus absolutely vital. Incorrect position of the tube can be fatal through loss of the airway or through barotrauma of the airway and lungs possibly leading to cardiac arrest. The mid-tracheal point of the trachea is the perfect place for an intra-tracheal tube to be to guarantee ventilatory support without problems for neonates and children. Supra-sternal palpation of the tube tip (SSTTP) is a method validated in newborns only, which has a very high accuracy rate in placing the tube-tip at the mid-tracheal point. In addition, it is easy to learn and without side effects. In infants and children, SSTTP is widely used in Switzerland although never validated in a controlled trial.

Objective:

To validate supra-sternal palpation of the endo-tracheal tube tip as a valuable measure to correctly determine the depth of intubation in infants from one month of age to children up to eight years of age, when correct depth of the tube-tip is defined as tube-tip being within plus/minus 0.25cm of the line between the medial points of the claviculae (IMP) for infants and within plus/mius 0.25 respectively plus/mius 0.38cm for toddlers and children.

Hypothesis:

Supra-sternal Tube Tip Palpation (SSTTP) is a valid and easy to perform measure to identify the correct depth of intubation after oral or nasal tracheal intubation in infants, toddlers and children. Correct depth is defined as tube tip placed within plus/minus 0.25cm of the IMP for infants and within plus/minus 0.25 respectively plus/minus 0.38cm for toddlers and children.

Study design and methods:

Sixty-four toddlers and children and 18 infants will be enrolled into the study. Three Respiratory Therapists (RT) from the Pediatric Intensive Care Unit (PICU) will be trained in SSTTP before the start of the study. Successful training of the RTs will be confirmed by x-ray before final qualification as "Expert in SSTTP". All patients with an intubation requiring a post-manipulation x-ray in the PICU at CHEO will be enrolled into the study. No randomization will be necessary; all infants and children in need of an intubation will be enrolled into the study. Potential patients will be excluded if there is presence of anatomical malformation or any other reason that would prevent accurate SSTTP, or if there is no Expert in SSTTP available. The location of the tip of the tube after SSTTP will be measured on standard post-intubation x-rays by a radiologist. The tube-tip location difference will be calculated as the difference between the actual tube-tip location and the IMP.

ELIGIBILITY:
Inclusion Criteria:

* "Primary intubations":

  * All infants and children from 1 month of age up to the end of the seventh year of life, who are being intubated for medical reasons on the pediatric intensive care unit (PICU) at the Children's hospital of Eastern Ontario.
* "Secondary intubations":

  * All infants and children from 1 month of age up to the end of the seventh year of life already intubated in the PICU at the Children's Hospital of Eastern Ontario, who's tube needs to be exchanged, who's tube needs to be repositioned according a previous x-ray or who's tube needs any other manipulation requiring a post-manipulation chest x-ray.

Exclusion Criteria:

* "Primary, peracute intubations". Intubations required at once or within a few minutes.
* Anatomical malformation of the child's or infant's airway, lungs or neck.
* Tracheostoma, history of tracheotomy, jugular scars or any other reason that might prevent accurate supra-sternal palpation.
* After placement of the tube according to supra-sternal palpation, any difficulties ventilating the patient or endo-bronchial intubation as per auscultation will lead to placement of the tube according to previously used criteria. The case will be described but the patient excluded from determination of the tube tip placement with x-ray.
* Any case when the study procedures had to be discontinued because the treating physician or RT felt that care could be disrupted by virtue of the study procedures. The case will be described but the patient excluded from determination of the tube tip placement with x-ray.
* Unavailability of an expert in SSTTP at the time point of needed intubation.
* For ethical reasons, we will exclude patients who we know will have a detrimental outcome despite intubation.

Ages: 1 Month to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-12 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Tube Placement with SSTTP | acute

SECONDARY OUTCOMES:
Ease of performing SSTTP | acute

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Schwarz, M.D., Dr. med., Principal Investigator — Department of Anesthesia, Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada